CLINICAL TRIAL: NCT02919553
Title: Modified Wet Suction Versus Capillary Techniques for EUS Guided Fine Needle Aspiration and Biopsy of Solid Lesions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: decided not to proceed with study at this time
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Alexander Jahng, MD, Gastroenterology attending, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 5160355
Record Dates: First submitted 2016-08-28; First posted 2016-09-29 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Pancreatic Cancer; Stomach Neoplasms
Keywords: endoscopic ultrasound; wet-suction technique; capillary technique; fine needle aspiration; fine needle biopsy
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified wet-suction technique (Experimental): Patients in this arm will undergo the modified wet-suction technique. Details in the study description section. After sufficient sampling of the lesion, the needle will be removed and the specimen will be collected.
  Interventions: Procedure: modified wet-suction technique
- Capillary "slow pull" technique (Active Comparator): Patients in this arm will undergo the Capillary "slow pull" technique which will include moving the needle to-and-fro into the lesion. Subsequently the needle will be removed and the specimen will be collected.
  Interventions: Procedure: Capillary "slow pull" technique

INTERVENTIONS:
Procedure: modified wet-suction technique — Normal saline will be present in this needle, and once in the lesion of interest the suction will be re-established and the needle will be moved in a to-and-fro motion to collect the sample of interest. Then the sample will be collected.
  Arms: modified wet-suction technique
Procedure: Capillary "slow pull" technique — The needle will be introduced into the lesion of interest and using the to-and-fro motion, collect the sample. The needle will then be withdrawn and the sample will then be collected.
  Arms: Capillary "slow pull" technique

SUMMARY:
The purpose of the study is to compare two particular techniques of tissue (capillary vs wet-suction techniques) sampling during endoscopic ultrasound guided fine needle aspiration/biopsy (EUS-FNA/FNB) of a solid lesion to determine the diagnostic yield and procedure logistics (e.g. procedure time).

DETAILED DESCRIPTION:
All adult patients who are undergoing EUS for solid lesions at Loma Linda University Health gastroenterology lab. These patients will be recruited at the time preceding their endoscopy in the Gastroenterology lab. They will be explained the goals, randomization, and interventions of the study. The collected patient information, as well as the steps to safeguard the information, will be explained.

Patients will be randomly assigned to capillary or wet-suction techniques arms according to computerized randomization program that has already been generated.

All patients will undergo routine EUS under possible moderate sedation or general anesthesia, with FNA/FNB. Cook Pro-core 22 gauge needle will be used for all the procedures. For each lesion undergoing FNA/FNB procedure, a total of 4 passes will be made using the selected technique.

The research aspect differentiates the method of tissue acquisition: modified wet-suction technique versus the "slow pull" capillary technique.

For the modified wet-suction technique:

1. The stylet will be removed at the onset of procedure. It will not be used unless it is necessary to de-clog the needle. Each de-clogging, if necessary, will be noted.
2. 10 mL suction syringe filled with saline will be used first to prime the needle until there is about 5 mL of saline left within the syringe
3. Then the plunger will be withdrawn against the locked three-way stopcock to establish vacuum. After this initial step, syringe with saline will not be removed for the entirety of the procedure unless technical issues arise, e.g. de-clogging.
4. Once the needle is introduced into the lesion of interest, the suction will be re-established by opening the three-way stopcock.
5. 10-20 to-and-fro needle motions will be done, emphasizing the edges of the lesion with fanning.
6. At the termination of each pass, the three-way stopcock will be closed prior to withdrawal of the needle from the lesion, to prevent suction of the specimen into the syringe itself.
7. Prior to steps to collect the specimen, the vacuum will be released, and after which the three-way stopcock will be turned to the open position.
8. Then the syringe plunger will then be pushed to collect the first drop of the specimen onto the glass slide for smear (thus making two glass smears for each pass, which will then be preserved into alcohol), and then the rest will be expunged onto the formalin for cell block.
9. Then the vacuum will be re-established as noted in step 3, ready for further needle passes.
10. For the first three passes, collection for both smear and the cell block will be done. For the last pass, all specimens will be collected on to the same cell block. Thus 6 total slides (which will be numbered or lettered consecutively for identification), and 1 formalin jar for cell block will be made for each patient/lesion.
11. Again, unless technical issues arise, the syringe will not be removed once initial priming is done and vacuum is established. Any technical issues will be noted within the procedure report.

For the capillary "slow pull" technique:

1. With the stylet slightly pulled back, the needle will be introduced into the lesion of interest, at which time the stylet will be pushed in to expunge any contaminating material.
2. The stylet will be slowly withdrawn by an assistant until completely removed.
3. 10-20 to-and-fro needle motions will be done, emphasizing the edges of the lesion with fanning.
4. After removal of the needle from the lesion, the stylet will be re-inserted. The first drop of will be collected for tissue smear, while the rest will be expunged first by stylet, saline, then air into formalin jar for cell block.
5. Stylet will then be re-introduced, ready for further passes.
6. For the first three passes, collection for both smear and the cell block will be done. For the last pass, all specimens will be collected on to the same cell block. Thus 6 total slides (which will be numbered or lettered consecutively for identification), and 1 formalin jar for cell block will be made for each patient/lesion.

Specimen handling:

Tissue smears will undergo for Papanicolaou staining, and the tissues preserved in 10% formalin solution will be processed for cell block.

The subjects will follow up with the Gastroenterology Clinic and/or their referring doctor. Patient may be called or receive a letter regarding their pathology results and for further follow-up as needed, per routine

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (greater than 18 years of age) who are referred for EUS guided sampling of solid lesions.

Exclusion Criteria:

* Any patients with contraindication to EUS- fine-needle aspiration/fine-needle biopsy (FNA/B), including those on anti-platelet or on anti-coagulation therapy, or with congenital disorders.
* Patients with cystic lesions or submucosal lesions will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rate of core tissue acquisition adequate for histologic analysis. | 4 weeks

SECONDARY OUTCOMES:
Diagnostic yield will measure the percentage of tissue acquisition cases that matched up with the final diagnosis. | 4 weeks
  Each tissue acquisition histology with be compared to final histology or diagnosis and from this we can calculate a percentage of accurate tissue acquisition.
Procedure time | 4 weeks
Tissue smear and cell block cellularity will be graded along this scale: Cellularity, graded 0 = no cells, 1 = sparsely cellular, 2 = moderately cellular, and 3 = highly cellular. | 4 weeks
  Each case will tallied into each graded category as noted above: no cells, sparsely cellular, moderately cellular, highly cellular. From there a percentage from the total number can be ascertained, median and mode can be calculated. The different percentage between tissue smear and cell block can be evaluated.
Tissue smear and cell block will be assessed of blood contamination with this scale: graded 0 = free of contamination, 1 = contaminated, 2 = highly contaminated, with or without blood clots. | 4 weeks
  Each case will tallied into each graded category as noted above: 0 = free of contamination, 1 = contaminated, 2 = highly contaminated, with or without blood clots. From there a percentage from the total number can be ascertained, median and mode can be calculated. The different percentage between tissue smear and cell block can be evaluated.
Tissue smear and cell block will be assessed of insertion tissue contamination with this scale: graded 0 = free of contamination, 1 = contaminated, 2 = highly contaminated. | 4 weeks
  Each case will tallied into each graded category as noted above: 0 = free of contamination, 1 = contaminated, 2 = highly contaminated. From there a percentage from the total number can be ascertained, median and mode can be calculated. The different percentage between tissue smear and cell block can be evaluated.
Tissue smear and cell block will be assessed of diagnosis characteristic with this scale: 0 = not adequate, 1 = suspicious for particular etiology, 2 = diagnostic for etiology, e.g. cancer. | 4 weeks
  Each case will tallied into each graded category as noted above: 0 = not adequate, 1 = suspicious for particular etiology, 2 = diagnostic for etiology, e.g. cancer. From there a percentage from the total number can be ascertained, median and mode can be calculated. The different percentage between tissue smear and cell block can be evaluated.
Cell block will be assessed of presence of any core tissue with intact architecture with this scale: graded 0 = none, 1 = present but marginal adequacy, 2 = present and adequate. Dimensions of the largest core will be noted if possible. | 4 weeks
  Each case will tallied into each graded category as noted above: 0 = none, 1 = present but marginal adequacy, 2 = present and adequate. From there a percentage from the total number can be ascertained, median and mode can be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Jahng, M.D, Principal Investigator — Loma Linda Univ Medical gastroenterology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wani S, Muthusamy VR, Komanduri S. EUS-guided tissue acquisition: an evidence-based approach (with videos). Gastrointest Endosc. 2014 Dec;80(6):939-59.e7. doi: 10.1016/j.gie.2014.07.066. No abstract available. PMID 25434654
- [Background] Kim GH, Cho YK, Kim EY, Kim HK, Cho JW, Lee TH, Moon JS; Korean EUS Study Group. Comparison of 22-gauge aspiration needle with 22-gauge biopsy needle in endoscopic ultrasonography-guided subepithelial tumor sampling. Scand J Gastroenterol. 2014 Mar;49(3):347-54. doi: 10.3109/00365521.2013.867361. Epub 2013 Dec 11. PMID 24325591
- [Background] Krishnan K, Dalal S, Nayar R, Keswani RN, Keefer L, Komanduri S. Rapid on-site evaluation of endoscopic ultrasound core biopsy specimens has excellent specificity and positive predictive value for gastrointestinal lesions. Dig Dis Sci. 2013 Jul;58(7):2007-12. doi: 10.1007/s10620-013-2613-1. Epub 2013 Mar 17. PMID 23504350
- [Background] Keswani RN, Krishnan K, Wani S, Keefer L, Komanduri S. Addition of Endoscopic Ultrasound (EUS)-Guided Fine Needle Aspiration and On-Site Cytology to EUS-Guided Fine Needle Biopsy Increases Procedure Time but Not Diagnostic Accuracy. Clin Endosc. 2014 May;47(3):242-7. doi: 10.5946/ce.2014.47.3.242. Epub 2014 May 31. PMID 24944988
- [Background] Iwashita T, Nakai Y, Samarasena JB, Park DH, Zhang Z, Gu M, Lee JG, Chang KJ. High single-pass diagnostic yield of a new 25-gauge core biopsy needle for EUS-guided FNA biopsy in solid pancreatic lesions. Gastrointest Endosc. 2013 Jun;77(6):909-15. doi: 10.1016/j.gie.2013.01.001. Epub 2013 Feb 20. PMID 23433596
- [Background] Attam R, Arain MA, Bloechl SJ, Trikudanathan G, Munigala S, Bakman Y, Singh M, Wallace T, Henderson JB, Catalano MF, Guda NM. "Wet suction technique (WEST)": a novel way to enhance the quality of EUS-FNA aspirate. Results of a prospective, single-blind, randomized, controlled trial using a 22-gauge needle for EUS-FNA of solid lesions. Gastrointest Endosc. 2015;81(6):1401-7. doi: 10.1016/j.gie.2014.11.023. Epub 2015 Feb 27. PMID 25733127